CLINICAL TRIAL: NCT00939601
Title: Evaluating Behavioral Treatments to Improve Adherence to Continuous Positive Airway Pressure (CPAP) Therapy in People With Obstructive Sleep Apnea
Brief Title: Evaluating Behavioral Treatments to Improve Adherence to CPAP in People With Obstructive Sleep Apnea
Acronym: BREATHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other)
Responsible Party: Mark S. Aloia, PhD,, National Jewish Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R01HL067209 (NIH)
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Adherence to CPAP in Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; OSA; Adherence; CPAP; Cognition
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Motivational Enhancement Therapy (Active Comparator): MET will involve counseling sessions and phone calls, with a focus on building self-efficacy and providing personalized feedback on health and adherence patterns based on CPAP adherence monitoring.
  Interventions: Behavioral: Motivational Enhancement Therapy
- Educational Counseling (Active Comparator): ED will involve sessions and phone calls that include educational information, problem-solving, and adherence feedback from study staff.
  Interventions: Behavioral: Educational Counseling
- Standard Care (No Intervention)

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy
  Arms: Motivational Enhancement Therapy
Behavioral: Educational Counseling
  Arms: Educational Counseling

SUMMARY:
Obstructive sleep apnea (OSA) is a serious sleep disorder in which a person repeatedly stops breathing or experiences shallow breathing for short periods of time during sleep. The most common treatment for OSA is the use of a continuous positive airway pressure (CPAP) machine, but many people have trouble adhering to the treatment schedule. This study will evaluate the effectiveness of two behavioral therapy programs used in combination with CPAP for improving treatment adherence in people with OSA.

ELIGIBILITY:
Inclusion Criteria:

* OSA confirmed by polysomnography (PSG)
* CPAP is the prescribed form of treatment for OSA
* Judged by sleep physician to respond to CPAP

Exclusion Criteria:

* Apnea/hypoxia index (AHI) less than 15
* Diagnosis of another sleep disorder that causes arousals from sleep
* Past treatment for OSA
* Current substance abuse problem
* Diagnosis of a serious medical condition that would interfere with involvement in the study
* History of a major psychiatric disorder, other than depression
* Change in antidepressant medication in the 3 months before study entry

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

REFERENCES:
- [Derived] Aloia MS, Knoepke CE, Lee-Chiong T. The new local coverage determination criteria for adherence to positive airway pressure treatment: testing the limits? Chest. 2010 Oct;138(4):875-9. doi: 10.1378/chest.09-2237. Epub 2010 Mar 26. PMID 20348198